CLINICAL TRIAL: NCT03925675
Title: Differentiating Brain Tumor Recurrence From Treatment-Induced Necrosis Using 18F-Fluciclovine (Anti-18f-facbc) PET and Multiparametric MR Imaging
Brief Title: 18F-Fluciclovine PET and Multiparametric MR Imaging
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No subjects enrolled
Sponsor: Loma Linda University (Other)
Collaborators: Blue Earth Diagnostics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 5180227
Record Dates: First submitted 2019-04-19; First posted 2019-04-24 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Brain Tumor, Recurrent, Adult
MeSH Terms: conditions — Brain Neoplasms; Recurrence | interventions — fluciclovine F-18

STUDY DESIGN:
Intervention Model Description: Subject who agree to participate in this study prior to surgery and sign the consent document, will have the following procedures done:
  1. Axumin (fluciclovine-F18) PET/CT scan will be done to evaluate possible recurrence to help differentiate scar (fake recurrence) from true tumor recurrence, which could be at any time point after initial surgery.
  2. Standard of care imaging surveillance will be done after initial tumor surgery
  3. Standard of care surgery will include the removal of the tumor.
  Tumor sample will then be analyzed and compared to the imaging (comparison of MRI, MRSI, and Axumin (fluciclovine-F18) imaging) results to determine an accurate diagnosis and location of tumor in the body.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Axumin (fluciclovine-F18) PET/CT scan (Experimental): Axumin (fluciclovine-F18) PET/CT scan to evaluate possible glioma recurrence to help differentiate scar (fake recurrence) from true tumor recurrence
  Interventions: Drug: PET/CT with F-Fluciclovine (Axumin)

INTERVENTIONS:
Drug: PET/CT with F-Fluciclovine (Axumin) — Comparison between PET/CT, MRI / MRS imaging, and biopsy histopathology. Data from each modality will be analyzed separately as described above to determine tumor recurrence and/or presence of radiation changes. Different metabolic profiles measured in areas of imaging changes and depicted by PET imaging will be characterized. Biopsy locations from stereotactic MRI data will be co-localized with PET/CT and MRSI to correlate biopsy histopathology with MRI+, MRSI+ and PET+ lesion data.
  Other Names: Axumin

SUMMARY:
The purpose of the study is to investigate the use of the investigational agent Axumin (fluciclovine-F18) with PET/CT imaging in combination with standard MR imaging to detect remaining or recurrent brain tumor.

DETAILED DESCRIPTION:
Methods:

Patients with recurrent enhancing mass on MRI in the side of a diagnosed and treated high grade glioma or metastatic brain tumor and consenting to study protocol will undergo 18F-Fluciclovine PET/CT imaging once prior to surgery for brain tumor recurrence. Surgery for recurrent brain tumor will follow standard of care treatment that includes either biopsy of the region or interest or as complete as possible tumor resection followed by histopathological analysis. Outcome evaluation will be analysis of tumor histology and imaging results, comparison of MRI, MRSI, and 18F-Fluciclovine imaging and relationship of imaging findings with histopathology and anatomical location of recurrent tumor.

Study Objectives

1. In this study, we will investigate the potential of 18F-fluciclovine to aid the visualization of residual or recurrent gliomas as depicted by 18F-Fluciclovine PET imaging compared to standard MRI sequences [T1 weighted imaging (T1WI) with contrast, diffusion weighted imaging (DWI), perfusion weighted imaging (PWI), T2 weighted fluid attenuated inversion recovery (T2 FLAIR)] using 3D image fusion.
2. To assess the residual or recurrent of glioma as depicted by 3D short echo time MR spectroscopic imaging (MRSI) using metabolic tumor markers such as elevated choline, myo-Inositol and lipids and reduced N-acetyl-aspartate (NAA) compared to standard MRI sequences (T1WI with contrast, PWI, T2 FLAIR) using 3D image fusion before neurosurgical intervention.
3. To spatially register the residual or recurrent glioma as depicted by 18F-Fluciclovine PET imaging with MR T1WI, DWI, PWI, and 3D MRSI to a) quantitate (SUVmax, SUVmean, ADCmean, rCBV, Cho, NAA, lipids, Cho/Cr, Cho/NAA) and correlate areas of PET+, T1WI+ and MRSI+ areas and b) characterize different metabolic profiles measured with MRSI in areas of glioma infiltration depicted by PET imaging and MRI.
4. Biopsy and pathology confirmation of tumor vs treatment-induced necrosis in spatially registered areas of interest will be performed.

Safety analysis Although 18F-Axumin™ is an FDA approved PET imaging agent for biological recurrent prostate cancer with extensive safety and toxicity data already documented, all patients will be monitored closely for adverse reactions after administration.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with prior histological confirmation of glioma or metastatic brain tumor evaluated for tumor recurrence or radiation changes after initial treatment of surgery, external beam radiation and / or chemotherapy with temozolamide.
2. Male and female
3. Ages 18 or greater

Exclusion Criteria:

1. Patient diagnosis with glioma or metastatic brain tumor but prior to surgery, external beam radiation and /or chemotherapy
2. Women who were pregnant, breast feeding, or possibly pregnant.
3. Patients with hepatic or renal dysfunction.
4. Patients with MRI contraindications (i.e. pacemakers, non-MR compatible devices).
5. Patients with a history of drug hypersensitivity to 18F-Fluciclovine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-08-24 (Estimated); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
18F-Fluciclovine | 2 years
  Investigate the potential of 18F-fluciclovine to aid the visualization of residual or recurrent gliomas as depicted by 18F-Fluciclovine PET imaging compared to standard MRI sequences [T1 weighted imaging (T1WI) with contrast, diffusion weighted imaging (DWI), perfusion weighted imaging (PWI), T2 weighted fluid attenuated inversion recovery (T2 FLAIR)] using 3D image fusion.
3D short echo time MR spectroscopic imaging (MRSI) | 2 years
  Using metabolic tumor markers such as elevated choline, myo-Inositol and lipids and reduced N-acetyl-aspartate (NAA) compared to standard MRI sequences (T1WI with contrast, PWI, T2 FLAIR) using 3D image fusion before neurosurgical intervention.
18F-Fluciclovine PET imaging with MR T1WI, DWI, PWI, and 3D MRSI | 2 years
  Quantitate (SUVmax, SUVmean, ADCmean, rCBV, Cho, NAA, lipids, Cho/Cr, Cho/NAA) and correlate areas of PET+, T1WI+ and MRSI+ areas and b) characterize different metabolic profiles measured with MRSI in areas of glioma infiltration depicted by PET imaging and MRI.
Biopsy and pathology | 2 years
  Confirmation of tumor vs treatment-induced necrosis in spatially registered areas of interest will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Warren Boling, MD, Principal Investigator — Loma Linda University Medical Center
Locations (1):
- Loma Linda University Cancer Center, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kotecha R, Aboian M, Nabavizadeh SA, Parent EE, Trifiletti DM, Chao ST. Letter regarding "Contribution of PET imaging to radiotherapy planning and monitoring in glioma patients-a report of the PET/RANO group": 18F-fluciclovine and target volume delineation. Neuro Oncol. 2021 Aug 2;23(8):1408-1409. doi: 10.1093/neuonc/noab097. No abstract available. PMID 34081125